CLINICAL TRIAL: NCT00395044
Title: Gabapentin for Cannabis Withdrawal and Use
Brief Title: Gabapentin Treatment of Cannabis Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Scripps Research Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Barbara J. Mason, Professor, The Scripps Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DA020766-01; 5R21DA020766-01 (NIH)
Record Dates: First submitted 2006-11-01; First posted 2006-11-02 (Estimated); Results first posted 2017-02-10 (Actual); Last update posted 2017-02-10 (Actual); Status verified 2016-12

CONDITIONS: Cannabis Dependence
Keywords: Cannabis treatment; marijuana treatment
MeSH Terms: conditions — Marijuana Abuse | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gabapentin (Experimental): 1200 mg/daily of Gabapentin
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator): 1200mg/d of Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Gabapentin
  Arms: Gabapentin

SUMMARY:
This is a study to evaluate the efficacy of the medication gabapentin in treating persons with cannabis dependence.

DETAILED DESCRIPTION:
This is a 12-week, double blind, placebo controlled, dose ranging study to evaluate the efficacy of gabapentin in treating outpatients with cannabis dependence. Counseling and research assessments occur weekly throughout the 12-week treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age 18-65 with cannabis dependence
* Meets DSM-IV-TR criteria for Cannabis Dependence
* Smoked marijuana at least once a week in the 90 days prior to study participation
* Willing to attend 12 weekly study visits and 1 follow-up visit

Exclusion Criteria:

* Currently meets DSM-IV-TR criteria for dependence on illicit substances other than cannabis
* Significant medical disorders that will increase potential risk or interfere with study participation
* Women with childbearing potential who are pregnant, nursing, or refuse to use a reliable method of birth control
* Treatment with an investigational drug in the last month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J. Mason, Ph.D., Principal Investigator — The Scripps Research Institute- Pearson Center for Alcoholism and Addiction Research
Locations (1):
- The Scripps Research Institute, La Jolla, California, United States

REFERENCES:
- [Result] Mason BJ, Crean R, Goodell V, Light JM, Quello S, Shadan F, Buffkins K, Kyle M, Adusumalli M, Begovic A, Rao S. A proof-of-concept randomized controlled study of gabapentin: effects on cannabis use, withdrawal and executive function deficits in cannabis-dependent adults. Neuropsychopharmacology. 2012 Jun;37(7):1689-98. doi: 10.1038/npp.2012.14. Epub 2012 Feb 29. PMID 22373942

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 50 subjects were recruited. An initial phone screen was conducted followed by an in-person clinical screening and interview in the research laboratory.
Pre-assignment Details: Subjects were excluded from enrollment if they did not meet Inclusion criteria or if they met one or more of the Exclusion criteria.
Groups:
- Placebo: Matched Placebo
Period: Overall Study
Arm/Group | Gabapentin | Placebo
Started | 25 | 25
Completed | 7 | 11
Not Completed | 18 | 14

BASELINE CHARACTERISTICS:
Population: All subjects who received a randomization number and packet of medication at week 1 were included in primary and secondary outcomes
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin | Placebo | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (8.5) | 34.4 (10.8) | 33.9 (9.7)
Gender [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 23 | 21 | 44
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Change From Week 0 in Cannabis Use Using Urinary CN-THCCOOH Levels at Week 12
Description: Urinary THC/Cr ratio, also known as CN-THCCOOH (creatinine normalized tetrahydrocannabinol carboxylic acid), is a highly sensitive and specific quantitative analytic procedure to determine current marijuana metabolite levels in the urine as well as new marijuana use or abstinence. Gas chromatography-mass spectrometric levels of 11-nor-9-carboxy-9-THC (THC-COOH), the primary marijuana metabolite, are normalized to the urine creatinine (CN) concentration to reduce the variability of drug measurement attributable to urine dilution. Negative values indicate decreased use.
Time Frame: Week 0 and Week 12
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 25 | 25
ng/ml | -966.00 (1175.25) | -532.81 (422.15)
Statistical Analysis 1: Comparison: Gabapentin vs Placebo; Test type: Superiority or Other; p = .029, Mixed Models Analysis

2. Secondary Outcome: Change From Week 0 in Withdrawal Symptom Severity on the Marijuana Withdrawal Checklist (MWC) at Week 12
Description: The MWC is an instrument to assess the severity of frequently reported cannabis withdrawal symptoms. Each question on the measure is recorded as a severity rating between 0-3: 0=best outcome; 3=worst outcome. The severity rating of each question was averaged to obtain a single marijuana withdrawal severity score. Change = (Week 12 score - Week 0 score).
Time Frame: Week 0 and Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 25 | 25
units on a scale | 1.42 (1.13) | 2.12 (1.50)

3. Secondary Outcome: Change in Sleep Quality on the Pittsburgh Sleep Quality Index (PSQI) at Week 12
Description: The PSQI is an instrument to assess subjective sleep quality and disturbance. The range on the measure is from 0-21: 0=best outcome; 21=worst outcome. Change = (Week 12 score - Week 0 score).
Time Frame: Week 0 and Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 25 | 25
units on a scale | -4.27 (3.07) | -1.72 (2.80)

4. Secondary Outcome: Change From Week 0 in Mood on the Beck Depression Inventory (BDI-II) at Week 12
Description: The BDI-II is a self-rating of severity of depressive symptoms. The Total score range on the BDI-II is from 0-63; 0=best outcome; 63=worst outcome. Change = (Week 12 score - Week 0 score).
Time Frame: Week 0 and Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 25 | 25
units on a scale | 3.71 (1.98) | 5.22 (2.36)

5. Secondary Outcome: Change From Week 0 in Craving on the Marijuana Withdrawal Checklist Marijuana Craving Question at Week 12
Description: The Marijuana Craving question of the Marijuana Withdrawal Checklist assesses severity of craving to smoke marijuana. The craving question is rated on a scale of 0-3 where 0=best outcome (no symptoms) and 3=worst outcome (severe symptoms). Change = (Week 12 score - Week 0 score).
Time Frame: Week 0 and Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 25 | 25
units on a scale | -1.55 (.64) | -1.46 (.77)

6. Secondary Outcome: Change From Week 0 in Cannabis-related Problems on the Marijuana Problem Scale (MPS) at Week 12
Description: The MPS is an instrument to assess the incidence of physical, psychological, social, and functioning problems that can result from cannabis dependence. The Total score ranges from 0-38 where 0=best outcome and 38=worst outcome. Change = (Week 12 score - Week 0 score).
Time Frame: Week 0 and Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 25 | 25
units on a scale | -3.40 (2.07) | -4.90 (7.09)

7. Secondary Outcome: Change From Baseline in Cognitive Functioning Using the Delis-Kaplan Executive Function System (D-KEFS) at Week 4
Description: The D-KEFS is a testing battery designed to measure executive functioning, a critical component of participating in cognitive behavioral therapy used to treat marijuana dependence. Data were obtained from the D-KEFS test instruments completed at baseline and week 4, which included the Trail Making Test, Verbal Fluency Test, and Color-Word Interference Test. Scaled scores range from 1 (worst) to 19 (best). Change = (Week 4 score - Week 0 score). Positive values indicate increased executive functioning.
Time Frame: Week 0 and Week 4
Population: Cognitive testing was done in a subset of participants enrolled in the study, beginning with randomized subject #21 and continuing until the 50th subject was randomized. The number analyzed is the total number available for analysis that completed both the Baseline and Week 4 assessment.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 7 | 10
scores on a scale | .28 (.50) | -.20 (.31)

ADVERSE EVENTS:
Time Frame: 13 weeks, from baseline to week 13
Arm/Group | Gabapentin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 16/25 | 14/25
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gabapentin (N=25) | Placebo (N=25)
Headache (Nervous system disorders) | 4 | 6
Insomnia (Nervous system disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 3 | 1
Cold symptoms (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Fatigue (Nervous system disorders) | 1 | 2
Depression (Psychiatric disorders) | 2 | 1
Irritability (Psychiatric disorders) | 1 | 2
Allergic reaction (Immune system disorders) | 2 | 1
Appetite decrease (Metabolism and nutrition disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No